CLINICAL TRIAL: NCT05323929
Title: The Relationship Between Scar Formation and ESD Depth in Therapy for Gastric Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2021-0634
Record Dates: First submitted 2022-04-05; First posted 2022-04-12 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Early Gastric Cancer; Endoscopic Submucosal Dissection
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- deep ESD group (Experimental): Performed according to the ESD standard procedure, the depth of dissection includes the SM3 layer (submucosa 1/3 layer)
  Interventions: Procedure: ESD
- shallow ESD group (Experimental): Performed according to the ESD standard procedure, the depth of dissection does not include the SM3 layer (submucosa 1/3 layer)
  Interventions: Procedure: ESD

INTERVENTIONS:
Procedure: ESD — Endoscopic Submucosal Dissection for early gastric cancer

SUMMARY:
This study is a single-center, prospective, group-controlled clinical trial, aiming to clarify the relationship between the depth of dissection and scar formation in the treatment of early gastric cancer by ESD, and to provide high-quality evidence-based medicine for the treatment of early gastric cancer.

DETAILED DESCRIPTION:
This project intends to compare the scar size of ESD for early gastric cancer with different peeling depths, explore the relationship between ESD peeling depth, scar formation and gastric function, and clarify the differential impact of different peeling depths on the prognosis of patients. We plan to provide evidence for guidelines of early gastric cancer ESD treatment based on the related data. In further, the project show insight into a more effective clinical technique which profit patients better prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old and younger than 75 years old.
* Early gastric cancer (T1a stage) diagnosed by gastroscopy or ultrasonography, differentiated and no ulcer; or early gastric cancer (T1a stage), differentiated with ulcer, lesion diameter <3cm; or early gastric cancer (T1a stage), undifferentiated and No ulcer, lesion diameter <2cm.
* Pathological diagnosis of gastric cancer.
* No further treatment is required.
* Patients diagnosed for the first time without other serious gastrointestinal diseases.

Exclusion Criteria:

* Those who did not comply with the test requirements, obviously violated this protocol, or switched to other protocols in the middle of treatment.
* Advanced gastric cancer; or undifferentiated gastric cancer lesions > 2 cm in diameter; or differentiated gastric cancer with ulcer lesions > 3 cm in diameter.
* Coagulation disorders.
* Serious heart, liver, kidney and other diseases, can not tolerate ESD treatment.
* Patients with gastric cancer complications such as gastrointestinal bleeding and perforation that need emergency treatment.
* Patients with distant metastasis.
* Patients with other tumors, patients with a history of malignant tumors (except early carcinoma in situ.
* The patient himself requests to withdraw from the trial.
* The researcher believes that the patient is not suitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
scar area | 1 year
  the scar area after ESD for 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Xinliang Lu, professor, Study Director — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second affiliated hospital, school of medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Russo AE, Strong VE. Gastric Cancer Etiology and Management in Asia and the West. Annu Rev Med. 2019 Jan 27;70:353-367. doi: 10.1146/annurev-med-081117-043436. Epub 2018 Oct 24. PMID 30355265
- [Background] Tsukuma H, Oshima A, Narahara H, Morii T. Natural history of early gastric cancer: a non-concurrent, long term, follow up study. Gut. 2000 Nov;47(5):618-21. doi: 10.1136/gut.47.5.618. PMID 11034575
- [Background] Toyonaga T, Man-i M, East JE, Nishino E, Ono W, Hirooka T, Ueda C, Iwata Y, Sugiyama T, Dozaiku T, Hirooka T, Fujita T, Inokuchi H, Azuma T. 1,635 Endoscopic submucosal dissection cases in the esophagus, stomach, and colorectum: complication rates and long-term outcomes. Surg Endosc. 2013 Mar;27(3):1000-8. doi: 10.1007/s00464-012-2555-2. Epub 2012 Oct 6. PMID 23052530
- [Background] Ono H, Yao K, Fujishiro M, Oda I, Uedo N, Nimura S, Yahagi N, Iishi H, Oka M, Ajioka Y, Fujimoto K. Guidelines for endoscopic submucosal dissection and endoscopic mucosal resection for early gastric cancer (second edition). Dig Endosc. 2021 Jan;33(1):4-20. doi: 10.1111/den.13883. Epub 2020 Dec 9. PMID 33107115
- [Background] Chung IK, Lee JH, Lee SH, Kim SJ, Cho JY, Cho WY, Hwangbo Y, Keum BR, Park JJ, Chun HJ, Kim HJ, Kim JJ, Ji SR, Seol SY. Therapeutic outcomes in 1000 cases of endoscopic submucosal dissection for early gastric neoplasms: Korean ESD Study Group multicenter study. Gastrointest Endosc. 2009 Jun;69(7):1228-35. doi: 10.1016/j.gie.2008.09.027. Epub 2009 Feb 27. PMID 19249769